CLINICAL TRIAL: NCT01105806
Title: The Use of a CPR Video to Enhance Advance Care Planning in Advanced Upper Gastrointestinal Cancer Patients: A Randomized Controlled Pilot Tria
Brief Title: Cardiopulmonary Resuscitation (CPR) Video to Enhance Advance Care Planning in Advanced Upper Gastrointestinal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Massachusetts General Hospital (Other); Mount Sinai Hospital, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 10-043
Record Dates: First submitted 2010-04-14; First posted 2010-04-19 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Pancreas and Hepatobiliary Cancer Patients
Keywords: advance directive; CPR Intervention; Video; Narrative; 10-043
MeSH Terms: conditions — Narration | interventions — Cardiopulmonary Resuscitation; Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- cardiopulmonary resuscitation (CPR) video: This pilot study involves a two-arm parallel design comparing the effectiveness of a CPR video versus a CPR narrative script in advance directive (AD) completion over a 1 month time frame post intervention.
  Interventions: Behavioral: (CPR) video and questionnaires
- cardiopulmonary resuscitation (CPR) narrative script: This pilot study involves a two-arm parallel design comparing the effectiveness of a CPR video versus a CPR narrative in advance directive (AD) completion over a 1 month timeframe post intervention.
  Interventions: Behavioral: cardiopulmonary resuscitation (CPR) narrative script and questionnaires

INTERVENTIONS:
Behavioral: (CPR) video and questionnaires — Baseline Assessments (10 mins),Intervention:CPR video or script (5 mins) Post intervention assessments (10 mins), Longitudinal chart review follow-up (6 months)
  Groups: cardiopulmonary resuscitation (CPR) video
Behavioral: cardiopulmonary resuscitation (CPR) narrative script and questionnaires — Baseline Assessments (10 mins),Intervention:CPR video or script (5 mins) Post intervention assessments (10 mins), Longitudinal chart review follow-up (6 months)
  Groups: cardiopulmonary resuscitation (CPR) narrative script

SUMMARY:
Advance care planning involves thinking about choices if the patient becomes sick, and is important for everyone. It does not matter if the patients are ill or healthy. It is especially important for people who have diseases that cannot be cured. It allows people to make sure their wishes are respected if they become very sick or are dying. Thinking about these issues can be upsetting. But, for many people, it is helpful. This type of discussion can help the family learn what the patient may want but cannot tell them when these decisions need to be made

ELIGIBILITY:
Inclusion Criteria:

* Primary pancreatic or hepatobiliary cancer (including ampullary carcinoma)as well as gastric and/or esophageal cancers, excluding neuroendocrine histology
* Progressive disease: Locally advanced or metastatic disease with progression on at least one course of treatment (surgery, radiation, or chemotherapy), or untreated patients unfit for therapy because of comorbidities or ECOG performance status >2, and finally, patients with ECOG performance status 2 -- patients must have discussed on at least one occasion with the treating investigator oncologist that their cancer cannot be cured
* In the estimation of the treating physician investigator, life expectancy ≤ 1 year
* Known to a GI medical oncology MSKCC clinic: Patients who have already established a relationship with a GI medical oncologist (who is an investigator on this protocol) after at least one new visit in the clinic (or as an in-patient), have MSKCC pathologist confirmed cancer of an above histology, and express an initial intent to be followed primarily at MSKCC
* English speaking*
* Able to provide informed consent
* Age greater than or equal to 18 years
* Do not have an advance directive or living will * English is the validated language in one of the study tools, and the language in which information is communicated in the narrative and video.

Exclusion Criteria:

* Short Portable Mental Status Questionnaire (SPMSQ) score of less than "intact mental functioning" (3 or more errors). SPMSQ in appendix.
* Any patient psychological state deemed by the treating physician to pose any risk of psychological harm by issues raised in a discussion of the trial, or in its testing procedures. Any subject who may become upset during any aspect or discussion of the study will be offered counseling services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the MSKCC GI medical oncology group of listed study investigators, and as above, 18 years of age or older with no advance directive completed, and will be English speaking, due to the study tools being based in English.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To document advance directive (AD)completion | 1 month post-test

SECONDARY OUTCOMES:
To assess patient uncertainty about, knowledge of, and preference for CPR. | pre and post randomization
To longitudinally follow discussions about ADs and nature of hospitalizations | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Reilly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm